CLINICAL TRIAL: NCT06270901
Title: Acute Effects of Legume-enriched Meals Compared to Western Diet Meals on Postprandial Metabolic Response in Women and Men At Increased Risk of Cardiovascular and Neurodegenerative Diseases
Brief Title: Acute Effects of Legume-enriched Meals Compared to Western Diet Meals on Postprandial Metabolism in Participants with Increased Cardiometabolic Risk
Acronym: LeguPlan_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: Federal Ministry of Food and Agriculture (BMEL) (Unknown); Federal Office for Agriculture and Food (BLE) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sarah Egert, Sarah Egert, Prof PhD, University of Bonn
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BMEL: 2822EPS008
Record Dates: First submitted 2024-02-02; First posted 2024-02-21 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome
Keywords: postprandial metabolic events
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High Protein Planetary Health Diet (Experimental): High Protein Planetary Health Diet Meal: This meal contains 62 g of protein primarily from plant origin (particularly legumes)
  Interventions: Other: High Protein Planetary Health Diet
- Low Protein Planetary Health Diet (Experimental): Low Protein Planetary Health Diet Meal: This meal contains 36 g of protein from primarily plant origin (particularly legumes)
  Interventions: Other: Low Protein Planetary Health Diet
- High Protein Western Diet (Experimental): High Protein Western Diet Meal: This meal contains 62 g of protein primarily form animal origin
  Interventions: Other: High Protein Western Diet
- Low Protein Western Diet (Experimental): Low Protein Western Diet Meal: This meal contains 36 g of protein primarily from animal origin
  Interventions: Other: Low Protein Western Diet

INTERVENTIONS:
Other: High Protein Planetary Health Diet — Planetary Health Diet Meal with 62 g of protein primarily from plant origin
  Arms: High Protein Planetary Health Diet
Other: Low Protein Planetary Health Diet — Planetary Health Diet Meal with 36 g of protein primarily from plant origin
  Arms: Low Protein Planetary Health Diet
Other: High Protein Western Diet — Western Diet Meal with 62 g of protein primarily from animal origin
  Arms: High Protein Western Diet
Other: Low Protein Western Diet — Western Diet Meal with 36 g of protein primarily from animal origin
  Arms: Low Protein Western Diet

SUMMARY:
The aim of the study is to investigate the postprandial effects of legume-enriched meals compared to Western Diet meals on postprandial metabolism. In this context, older adults with increased risk for cardiometabolic diseases consume 4 mixed meals with 36 g or 62 g of protein either designed according to the Planetary Health Diet with legumes as primary protein source or the Western Diet with animal foods as primary protein source, in a randomized order. In a postprandial observation period of 6 hours, parameters of lipid metabolism, glucose and insulin metabolism, amino acid profile, as well as markers of inflammation and vascular function are analysed. Furthermore, neuropsychological parameters and satiety-associated hormones are investigated.

DETAILED DESCRIPTION:
In a randomized crossover design, 30 older men and women with increased risk for cardiometabolic diseases consume 4 mixed meals, which differ in dietary pattern, protein source and protein quantity. Two meals are designed according to the Planetary Health Diet with legumes as primary protein source whereas the other two meals are designed according to the Western Diet with animal food as primary protein source. Two meals are designed as high protein meals (62 g of protein) and two meals are designed as low protein meals (36 g of Protein). Therefore, participants consume 4 different test meals, a Low and a High Protein Western Diet Meal and a Low and a High Protein Planetary Health Diet Meal in a randomized order. During a postprandial observation period of 6 hours, parameters of lipid metabolism (e.g., plasma triglycerides), glucose metabolism (e.g., plasma glucose, serum insulin), as well as markers of inflammation (e.g., IL-6) and vascular function (e.g., pulse wave velocity) are analysed. Furthermore, amino acid profile, neuropsychologic parameters (e.g., appetite) and satiety-associated hormones (e.g., Ghrelin) are investigated. Each intervention will be separated by a washout period of approximately 14 days.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* Non-smoking
* BMI: 27 - 34,9 kg/m2
* Waist circumference (women ≥ 80 cm, men ≥ 94 cm)
* Systolic blood pressure: ≥ 120 mmHg, diastolic blood pressure: ≥ 80 mmHg
* At least one of the following criteria
* Fasting triglycerides in serum: ≥ 150 mg/dL
* Fasting HDL-Cholesterol in serum: women < 50 mg/dl, men < 40 mg/dL
* Fasting C-reactive protein in serum: ≥ 2 mg/L
* Fasting glucose in plasma: ≥ 100 mg/dL

Exclusion Criteria:

* food intolerances and allergies (especially to legumes)
* Smoking
* malabsorption syndromes
* thyroid diseases
* impaired renal function
* chronic liver disease
* heart failure
* myocardial infarction
* insulin-dependent diabetes mellitus
* chronic inflammatory diseases
* tumors
* anemia
* immunosuppression
* intake of supplements (e.g., fish oil)
* Participation in another study
* other exclusion criteria at the discretion of the physician/ investigator

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Parameters of lipid metabolism in blood | Postprandial period of 6 hours (T=0, 1, 2, 3, 4, 6 hours)
  Triglycerides (mg/dL)

SECONDARY OUTCOMES:
Parameters of lipid metabolism in blood | Postprandial period of 6 hours (T=0, 1, 2, 3, 4, 6 hours)
  Total cholesterol (mg/dL)
Parameters of lipid metabolism in blood | Postprandial period of 6 hours (T=0, 1, 2, 3, 4, 6 hours)
  LDL cholesterol (mg/dL)
Parameters of lipid metabolism in blood | Postprandial period of 6 hours (T=0, 1, 2, 3, 4, 6 hours)
  HDL cholesterol (mg/dL)
Parameters of lipid metabolism in blood | Postprandial period of 6 hours (T=0, 1, 2, 3, 4, 6 hours)
  Free fatty acids (mmol/L)
Parameters of glucose metabolism in blood | Postprandial period of 6 hours (T=0, 0.5, 1, 1.5, 2, 3, 4, 6 hours)
  Glucose (mg/dL)
Parameters of glucose metabolism in blood | Postprandial period of 6 hours (T=0, 0.5, 1, 1.5, 2, 3, 4, 6 hours)
  Insulin (nmol/L)
Parameters of glucose metabolism in blood | Postprandial period of 6 hours (T=0, 0.5, 1, 1.5, 2, 3, 4, 6 hours)
  cPeptide (pg/mL)
Parameters of glucose metabolism in blood | Postprandial period of 6 hours (T= 0, 1, 2, 3, 4, 6 hours)
  GLP-1 (pg/mL)
Parameters of glucose metabolism in blood | Postprandial period of 6 hours (T= 0, 1, 2, 3, 4, 6 hours)
  Glucagon (pg/mL)
Blood amino acid profile | Postprandial period of 6 hours (T= 0, 1, 2, 3, 4, 6 hours)
  Amino acid profile in blood (nmol/mL)
Blood urea | Postprandial period of 6 hours (T=0, 1, 2, 3, 4, 6 hours)
  Urea in blood (mg/dL)
Uric acid in blood | Postprandial period of 6 hours (T=0, 1, 2, 3, 4, 6 hours)
  Uric acid in blood (mg/dL)
Parameters of hunger and satiety in blood | Postprandial period of 6 hours (T= 0, 1, 2, 3, 4, 6 hours)
  e.g. Ghrelin (pg/mL)
Parameters of endothelial function in blood | Postprandial period of 6 hours (T= 0, 1, 2, 3, 4, 6 hours)
  e.g. ADMA (µmo/L)
Parameters of inflammation in blood | Postprandial period of 6 hours (T= 0, 1, 2, 3, 4, 6 hours)
  e.g. IL-6 (pg/mL)
Endothelial function | Postprandial period of 6 hours (T=0, 2, 4, 6 hours)
  e.g. pulse wave velocity (m/s)
Neuropsychological parameters | Postprandial period of 6 hours (T=0, 0.5, 1, 1.5, 2, 3, 4, 5, 6 hours)
  Assessment of hunger and satiety via a visual analogue scale (e.g. 0 = not hungry at all to 10 = very hungry)
Neuropsychological parameters | Postprandial period of 4.5 hours (T= 0, 1.5, 3, 4.5 hours)
  Assessment of attention via questionnaire (paper pencil test, e.g. higher amount of marked target items = higher attention, maximum points 640 = every target items marked correctly, minimum points: 0 = no target items marked or only wrong items marked)
Neuropsychological parameters | Postprandial period of 6 hours (T=0.5, 3, 6 hours)
  Assessment of memory via questionnaire (paper pencil, e.g. higher reproduction of memorised visual and verbal information = better memory; visual part: maximum points: 31 = all visual information memorised, minimum points: 0 = no visual information memorised; verbal part: maximum points: 24 = all verbal information memorised, minimum points: 0 = no verbal information memorised)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn, Institute of Nutritional and Food Sciences, Nutrition Physiology, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No